CLINICAL TRIAL: NCT00558402
Title: Meditation for Alzheimer Caregivers: Stress & Physiology
Brief Title: Meditation or Education for Alzheimer Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Barry S. Oken, MD, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00002226
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Caregivers; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Meditation; Mindfulness-Based Stress Reduction; Educational Status; Caregivers; Respite Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Meditation class, 90min/week for 8 weeks, with home assignments, adapted from MBCT program
  Interventions: Behavioral: Meditation
- 2 (Active Comparator): Education
  Interventions: Behavioral: Education
- 3 (Active Comparator): Respite care only, 90 mins per week for 8 weeks
  Interventions: Behavioral: Respite only

INTERVENTIONS:
Behavioral: Meditation — meditation class 1/week for 8 weeks
  Other Names: Mindfulness Based Stress Reduction
  Arms: 1
Behavioral: Education — Education class, 90 min per week for 8 weeks along with home assignments based on Powerful Tools for Caregivers
  Other Names: Powerful Tools for Caregivers
  Arms: 2
Behavioral: Respite only — Respite care 90 mins per week for 8 weeks
  Other Names: Respite care
  Arms: 3

SUMMARY:
The goal is to determine how 6-week stress reduction techniques may decrease stress in primary caregivers of people with Alzheimer's disease. The 3 intervention programs are meditation, education, and respite care. There will be approximately 108 subjects over 3 years. Subjects will have a screening session over the phone to see if they are eligible (50-85 years old, spending at least 12 hours per week caring for a close relative with Alzheimer's disease, willing to be in any of the 3 groups, and without any very serious medical problem). The subjects will have 3 testing sessions, 1 before classes/respite and 2 after classes are over, each lasting about 3 hours. The classes are taught in a one-on-one setting, and they are 50 minutes per week for 6 weeks. Respite care is provided for the person with Alzheimer's disease in all the groups. Measurements include people's ratings of stress, psychological testing, and biological measurements of stress, including the following: saliva, blood, and urine collection; waist-to-hip ratio; weight; blood pressure; heart rate; respiration; reaction time task; voice recordings; electrocardiogram; electroencephalogram; and electro dermal activity.

DETAILED DESCRIPTION:
Stress has a negative effect on many aspects of health. Older adults may be particularly sensitive to adverse effects of stress because of lower physiologic reserves and coexistence of other health problems. Since mind-body interventions may be most effective in conditions associated with psychological stress, this research will evaluate the effectiveness of a mind-body intervention in seniors who have a significant stress: being the primary caregiver for a person with dementia (PWD) secondary to Alzheimer's disease. The well-being of this large and growing group of Americans is a significant public health issue. We plan to study a Mindfulness Based Cognitive Therapy (MBCT) program for caregivers of a PWD in a randomized 3-arm intervention trial. There are two comparison groups: an education group and a pragmatic, respite only group. The two active interventions, MBCT and education, also include identical respite care for the PWD to allow the caregiver to attend the classes. Each intervention will last 6 weeks, and consist of one 50 minute class and/or or 2-3 hours of respite per week along. Homework for the two groups in the classes will consist of home meditation practice for the MBCT group and development of an action plan and reading for the education group. Outcome measures will be assessed at 8 weeks and at 20 weeks (immediately and 12 weeks after the intervention class has been completed). Our primary outcome measure will be a self-rated measure of caregiver stress. There are a number of secondary outcome measures representing biomarkers of stress including: salivary cortisols measured over the day to include the awakening response and trough levels; inflammatory markers; and electrophysiologic markers. Other secondary outcome measures include self-efficacy, health-related quality of life, mood, and cognitive function. We will use several measures to predict response to MBCT and education in an aptitude by treatment interaction analysis. These measures include the personality trait absorption, emotion-based versus problem-based coping, and expectancy of improvement from each intervention. We will also use the 24-hour acquisition device to evaluate the ability of subjects randomized to MBCT to induce physiologic changes during self-reported mindfulness meditation and relate the magnitude of these changes to improvements in outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 50-85 year olds who are the primary caregiver of someone with Alzheimer disease (family member or other close relationship)

Exclusion Criteria:

* cognitively impaired
* unstable medical problems
* untreated significant depression
* taking CNS-active medications that have not been stable for 2 months
* significant visual impairment (acuity worse than 20/50 OU)
* experience with meditation classes of with Powerful Tools for Caregivers classes
* not have significant baseline stress
* evidence on history of certain significant neurological diseases
* unwilling to accept randomization or to commit to attending classes and practicing the interventions

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Caregiver stress (Revised Memory and Behavior Problems Checklist) | 8 and 20 weeks

SECONDARY OUTCOMES:
5-Facet Mindfulness Questionnaire | 0, 8 and 20 weeks
  This self-report questionnaire measures different aspects of mindfulness
Perceived Self-Efficacy | Measured 0, 8, and 16 Weeks
  The General Perceived Self-Efficacy Scale developed by Schwarzer and Jerusalem in 1995 contains 10 items asking about sense of control.
EEG measuring reaction time | Measured at 0, 8, and 16 weeks
  EEG is recorded during reaction time tests to measure attention

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Oken, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States